CLINICAL TRIAL: NCT02935192
Title: A Phase 3 Double Blinded, Randomized, Placebo- Controlled Study to Examine the Safety and Immunogenicity of a Seasonal Trivalent Split Inactivated Influenza Vaccine Produced by Institute Torlak in 18-65 Year Old Volunteers in Serbia
Brief Title: Phase 3 Trial of Serbian Seasonal Influenza Vaccine
Acronym: Torlak-300
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Virology, Vaccines and Sera, Torlak (Other)
Collaborators: PATH (Other); Comac Medical (Industry); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Torlak-300; VAC 053 (Other: PATH)
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Influenza
Keywords: seasonal influenza; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine Arm (Experimental): Seasonal trivalent split, inactivated influenza vaccine
  Interventions: Biological: Vaccine
- Placebo Arm (Placebo Comparator): Phosphate buffered saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Vaccine — Seasonal trivalent split, inactivated influenza vaccine 15 mcg hemagglutinin antigen (HA) of each of A/H1N1; A/H3N2 and B strains; 0.5 mL by IM injection
  Arms: Vaccine Arm
Other: Placebo — Phosphate buffered saline, 0.5 mL by IM injection
  Arms: Placebo Arm

SUMMARY:
A Phase 3, double-blind, randomized, placebo-controlled trial of a seasonal, trivalent, split, inactivated influenza vaccine produced by InstituteTorlak.

DETAILED DESCRIPTION:
This is a phase 3, double-blind, randomized, placebo- controlled trial with two groups of participants to receive seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or placebo (phosphate buffered saline). A total of about 480 healthy male and female adults 18 through 65 years of age; 320 participants will be randomized to receive vaccine and160 will receive placebo (a 2:1 ratio). At least 25% of the participants (N=120) will be >/= 45 years of age (80 vaccine and 40 placebo recipients).

Safety will be assessed in all participants through Day 91. Immunogenicity will be assessed in serum samples obtained at baseline and 21 days after vaccination in a subset of at least 100 individuals randomized to study vaccine and 50 placebo recipients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years on the day of screening/enrollment.
* Literate (by self-report) and willing to provide written informed consent.
* Able to attend all scheduled visits and to comply with all trial procedures.
* Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable under control or unchanged for the past three months. If medication is used to treat the condition, the medication dose must have been stable for at least one month preceding vaccination.

For female participants:

* Not breast feeding, non-pregnant (based on negative urine pregnancy test) and no plan to become pregnant up to Day 22.
* Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than one year must be willing to use effective contraceptive method to prevent pregnancy until three weeks (Day 22) after vaccination. Effective methods include intrauterine device, hormonal contraceptives (oral, injectable, patch, implant, ring) or double barrier contraceptives (condom or diaphragm with spermicide). Women with credible history of abstinence may be enrolled at the discretion of the investigator.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of influenza vaccine in the last 10 months.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 22 visit.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products prior to the Day 22 visit.
* Known or suspected congenital or acquired immunodeficiency.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, ≥ 0.5 mg per kg per day; topical steroids are allowed.)
* Unstable illness by history or physical examination that in the opinion of the investigator, might interfere with the conduct or results of the study or pose additional risk to the participant.
* Hypersensitivity after previous administration of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein or antibiotics.
* Bleeding disorder or receipt of anticoagulants in the three weeks preceding enrollment.
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause (self-report).
* Current alcohol or drug addiction that in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* History of Guillain-Barré Syndrome.
* Neoplastic disease or any hematologic malignancy. Allowed: localized skin or prostate cancer that is no longer being treated and is stable at the time of vaccination and participants who have a history of neoplastic disease and who have been disease free for ≥ 5 years.
* Any condition that, in the opinion of the investigator, would increase the health risk to the participant if he/she participates in the study, or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-01-08 (Actual); Study Completion 2017-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goran Stevanovic, MD, Study Chair — Clinical Center of Serbia, Clinic for Infectious and Tropical Diseases
Locations (6):
- Serbia (6):
  - Clinical Center of Serbia: Clinic for Infectious and Tropical Diseases, Belgrade
  - Clinical Center of Serbia: Clinic for Pulmonology, Belgrade
  - Institute for Students' Healthcare, Belgrade
  - Institute of Health Care of Workers of the Ministry of Internal Affairs, Belgrade
  - Jevremova Special gynecology hospital with maternity, Belgrade
  - General Hospital Vrsac, Vršac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevanovic G, Obradovic A, Ristic S, Petrovic D, Milenkovic B, Mitrovic D, Vignjevic SF, Ilic K, Stoiljkovic V, Lavadinovic L, Pelemis M, Petrovic S, Vidmanic A, Popovic O, Eremic N, Sparrow E, Torelli G, Socquet M, Holt R, Ilieva-Borisova Y, Tang Y, Scorza FB, Flores J, Rathi N. Safety and immunogenicity of a seasonal trivalent inactivated split influenza vaccine: a double blind, phase III randomized clinical trial in healthy Serbian adults. Ther Adv Vaccines Immunother. 2020 May 25;8:2515135520925336. doi: 10.1177/2515135520925336. eCollection 2020. PMID 32518891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 503 subjects were consented and screened from across 6 clinical trial sites located in Belgrade and Vrsac, Serbia. Of the 503 subjects screened, 23 subjects failed screening.
Pre-assignment Details: Twenty-three (23) subjects failed screening and were not assigned to a treatment group.
  An additional 8 subjects withdrew consent prior to receiving any study product.
Groups:
- Vaccine Arm: Trivalent seasonal influenza vaccine
Period: Overall Study
Arm/Group | Vaccine Arm | Placebo Arm
Started | 320 (312 subjects were included in the Full Protocol Analysis because 8 withdrew without getting product.) | 160 (156 subjects were included in the Full Protocol Analysis because 4 withdrew without getting product.)
Received Vaccine/Placebo | 312 | 156
Completed | 312 | 156
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Population: Participants enrolled and vaccinated without major protocol deviations
Groups:
- Vaccine: Seasonal trivalent split, inactivated influenza vaccine
  Seasonal Influenza Vaccine: Seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B); 0.5 mL by IM injection
- Placebo: Phosphate buffered saline
  Phosphate Buffered Saline: Phosphate buffered saline, 0.5 mL by IM injection
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 312 | 156 | 468
Age, Continuous [Mean (Full Range); unit: years] — Population: Each row represents a subpopulation of age range for the study (18-44 years; 45-65 years). Together these totals add up to the overall study population in each arm.
  years
    18-44 years: number analyzed (Participants) | 232 | 116 | 348
    18-44 years | 32.8 [18 to 44] | 32.0 [18 to 44] | 32.6 [18 to 44]
    45-65 years: number analyzed (Participants) | 80 | 40 | 120
    45-65 years | 54.7 [45 to 65] | 53.8 [45 to 63] | 54.4 [45 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 77 | 222
  Male | 167 | 79 | 246
Region of Enrollment [Number; unit: participants]
  Serbia | 312 | 156 | 468

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (Local & Systemic Reactogenicity)
Description: Number of participants experiencing one or more solicited local AEs, including redness /erythema, swelling / induration and pain
Time Frame: 30-minute post-vaccination period
Population: The analysis was conducted for subjects who were randomized and received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 312 | 156
Participants
  Hardness | 5 | 1
  Pain | 5 | 0
  Redness | 22 | 3
  Swelling | 1 | 0
  Tenderness | 2 | 0
  Temperature above 37 C | 0 | 0
  Chills | 0 | 0
  Headache | 0 | 0
  Joint aches | 0 | 0
  Muscle aches | 0 | 0
  Nausea | 0 | 0
  Tiredness | 1 | 0

2. Primary Outcome: Number of Participants With Solicited Local Adverse Events (Local Reactogenicity)
Description: Number of subjects reporting one or more solicited local reactions (redness/erythema, swelling/induration, pain, and tenderness) at the injection site post-vaccination with study vaccine or placebo
Time Frame: 5-day period (Days 1-5) post-vaccination
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 312 | 156
Participants
  Hardness | 29 | 0
  Pain | 160 | 17
  Redness | 40 | 3
  Swelling | 20 | 0
  Tenderness | 126 | 11

3. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (Systemic Reactogenicity)
Description: Number of subjects reporting one or more solicited systemic reactions (fever, fatigue/malaise, muscle aches, joint aches, chills, nausea, vomiting, and headache) post-vaccination with study vaccine or placebo.
Time Frame: 5-day period (Days 1-5) post-vaccination
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 312 | 156
Participants
  Chills | 11 | 1
  Headache | 47 | 19
  Joint Aches | 16 | 5
  Muscle Aches | 27 | 6
  Nausea | 18 | 6
  Temperature | 6 | 1
  Tiredness | 53 | 16

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited AEs occurring in 1% or more of study participants; includes events irrespective of causality
Time Frame: Within 21 days post vaccination
Population: Full analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 312 | 156
Participants
  Nasopharyngitis | 3 | 4
  Respiratory tract infection | 7 | 1
  Rhinitis | 3 | 3

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: Number of participants reporting one or more of all anticipated and unanticipated serious adverse events, grouped by organ system, with number and frequency of such events in each arm/group of the clinical study.
Time Frame: Over the entire study period (Day 91)
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 312 | 156
Participants
  Acute Lymphocytic Leukemia: Related | 0 | 0
  Acute Lymphocytic Leukemia: Not related | 1 | 0
  Acute Lymphocytic Leukemia: Not reporting this SAE | 311 | 156
  Varicocele: Related | 0 | 0
  Varicocele: Not related | 1 | 0
  Varicocele: Not reporting this SAE | 311 | 156

6. Primary Outcome: Number and Percentage of Seroconverted Subjects
Description: Seroconversion is defined as a serum HAI antibody titer meeting the following criteria:
  * Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day 22 of ≥1:40; or
  * Pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination measured on Day 22.
  Measured against each of the 3 antigens
Time Frame: Day 22
Population: Per Protocol (PP) Population:
  Immunogenicity was assessed in a subset of 151 participants (per-protocol population) with valid post-vaccination immunogenicity measures and no major protocol violations that were determined to potentially interfere with the immunogenicity assessment of the study vaccine. This was decided before unblinding.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 101 | 50
Participants
  Seroconversion to H1 | 91 | 1
  Seroconversion to H3 | 77 | 0
  Seroconversion to B | 52 | 9

7. Primary Outcome: Number and Percentage of Participants With a HAI Antibody Titer ≥1:40 (Seroprotection)
Description: Seroprotective Titers is considered as HAI antibody Titre ≥1:40; measured for each of the 3 antigens
Time Frame: Day 1 and Day 22
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 101 | 50
Participants
  Seroprotection to H1N1 : Day 1 | 24 | 21
  Seroprotection to H1N1 : Day 22 | 96 | 22
  Seroconversion to H3N2 : Day 1 | 7 | 3
  Seroconversion to H3N2 : Day 22 | 79 | 3
  Seroprotection to B : Day 1 | 53 | 18
  Seroprotection to B : Day 22 | 93 | 26

8. Primary Outcome: Geometric Mean Titers (GMTs) of Serum HAI Antibodies
Description: Serum HAI Antibodies GMTs Pre- (Day 1) and Post-vaccination (Day 22); measured for each of the 3 antigens
Time Frame: Day 1 and Day 22
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 101 | 50
Titer
  GMT to H1 : Day 1 | 15.0 [12.3 to 18.1] | 24.1 [16.9 to 34.5]
  GMT to H1 Day 22 | 336.3 [268.2 to 421.7] | 25.0 [17.7 to 35.2]
  GMT to H3 : Day 1 | 6.9 [6.0 to 7.8] | 8.0 [6.4 to 10.0]
  GMT to H3 : Day 22 | 88.4 [65.9 to 118.5] | 8.4 [6.6 to 10.5]
  GMT to B : Day 1 | 27.4 [21.6 to 34.8] | 21.9 [15.8 to 30.3]
  GMT to B : Day 22 | 103.5 [86.9 to 123.3] | 36.1 [26.7 to 48.7]

9. Primary Outcome: Geometric Mean Fold Rises (GMFRs) of Serum HAI Antibodies
Description: GMFR calculated as GMT for of Serum HAI Antibodies Post-vaccination/Pre-vaccination; measured for each of the 3 antigens
Time Frame: Day 1 and Day 22
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Vaccine Arm | Placebo Arm
Number analyzed (Participants) | 101 | 50
Titer
  GMFR for H1 | 22.5 [17.5 to 28.9] | 1.0 [0.9 to 1.2]
  GMFR for H3 | 12.9 [9.8 to 17.0] | 1.0 [1.0 to 1.1]
  GMFR for B | 3.8 [3.0 to 4.8] | 1.6 [1.3 to 2.1]

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Vaccine: Trivalent seasonal influenza vaccine
- Placebo: Phosphate buffered saline
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/312 | 0/156
Serious Adverse Events (participants affected / at risk) | 2/312 | 0/156
Other Adverse Events (participants affected / at risk) | 13/312 | 8/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=312) | Placebo (N=156)
Acute Lymphocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Varicocele (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=312) | Placebo (N=156)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4)
Respiratory tract infection (Infections and infestations) | 7 (7) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No